CLINICAL TRIAL: NCT04365712
Title: Piezoelectric Tools Versus Traditional Oscillating Saw for Distal Linear Osteotomy in Hallux Valgus Correction: a Prospective, Triple-blinded, Randomized Controlled Study.
Brief Title: Osteotomy of the 1st Metatarsal for Hallux Valgus Using Pneumatic Oscillating Saw or Piezoelectric Scalpel
Acronym: Piezo-Hallux
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0035857
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2020-04

CONDITIONS: Hallux Valgus
Keywords: Hallux valgus; Radiographic consolidation; Piezoelectric scalpel
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Intervention Model Description: 40 patients affected by hallux valgus were recruited, based on the listed inclusion and exclusion criteria; 20 underwent 1st metatarsal osteotomy treated with a piezoelectric tool (experimental group) and 20 underwent 1st metatarsal osteotomy with a traditional oscillating saw (control group). The patients were randomly allocated (1:1) in a Piezoelectric Group (PG) and in a Control Group (CG) utilizing sealed envelopes. The envelopes were prepared and shuffled by the same senior surgeon involved in the surgical procedures and drawn by a researcher not involved in the surgical procedures or the clinical and radiographic assessment.
  3 patients in PG (1 did not comply with the post-operative management and 2 missed the scheduled follow-up appointments) and 3 patients in CG (all patients discontinued from the evaluations) were lost to follow-up.
  Thus, 17 patients in each group were evaluated in the 1-year analysis, all treated according to their original assignment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patient did not know with which instrument the osteotomy had been performed.
  The radiologist who certifies the osteotomy radiographic healing did not know with which instrument the osteotomy had been performed.
  The clinical investigator who collected the evaluation questionnaires was not aware of the type of instruments used during the surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oscillating saw (Active Comparator): Patients treated for hallux valgus with 1st metatarsal osteotomy obtained by common oscillating saw
  Interventions: Device: Oscillating Saw
- Piezoelectric tool (Experimental): Patients treated for hallux valgus with 1st metatarsal osteotomy obtained by piezoelectric tool
  Interventions: Device: Piezoelectric tool

INTERVENTIONS:
Device: Piezoelectric tool
  Arms: Piezoelectric tool
Device: Oscillating Saw
  Arms: Oscillating saw

SUMMARY:
The main goal of the surgical correction of the hallux valgus is the morphological correction associated with the functional rebalancing of the first ray. The aim of this study was to show the efficacy of piezosurgery in performing distal linear osteotomy of the first metatarsal bone in hallux valgus correction, in terms of clinical and radiological outcomes at 1-year final follow up.

DETAILED DESCRIPTION:
This study was performed collecting pre-operative and post-operative data for all patients.

At the time of admission, the patients received and signed an Informed Consent to adhere to the Study Protocol. On this occasion, the patients were also given a summary scheme of the clinical and radiographic checks to which they would have undergone in case of adherence to the Study Protocol.

40 patients were included in the trial and were randomly allocated (1:1) in a Piezoelectric Group (PG) and in a Control Group (CG) (that provided for the use of a traditional oscillating saw) utilizing sealed envelopes. The envelopes were prepared and shuffled by the same senior surgeon involved in the surgical procedures and drawn by a researcher not involved in the surgical procedures or the clinical and radiographic assessment.

The patients were not aware of the instrument used during surgery. In both groups, patients were treated with the same surgical technique, a distal linear osteotomy of the first metatarsal bone (S.E.R.I. technique). Clinical and radiographic assessments were performed during the multiple follow-ups.

The final follow-up was at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Mild to moderate hallux valgus (Hallux valgus Angle <; 40° and Intermetatarsal Angle < 20°),
* No osteoarthritis or grade 1 osteoarthritis of the first metatarsophalangeal joint (MTPj) according to Regnauld grading

Exclusion Criteria:

* Stiffness of the first MTPj or osteoarthritis ≥ grade 2 according to Regnauld's classification
* Rheumatoid arthritis or other chronic inflammatory joint diseases
* Diabetes
* Neurological disorders
* Previous hallux valgus surgical corrections
* Hypermobility of the first MTPj as per congenital laxity syndromes.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-10-24 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
23/5000 Radiographic healing. Patients underwent several radiographic checks, pre-operatively and follow-ups, in order to analyze the healing changes in the osteotomy of 1 metatarsus | Preoperative, 21-35-50-70-90-180-360 days of follow up from the surgery
  The patients underwent radiographic control (foot in two projections under load) preoperatively and at 21-35-50-70-90-180-360 days of follow up from the surgery. The radiographs obtained were evaluated by an independent radiologist, always the same for the duration of the study, who was not aware of the type of instrument used during the surgery. His task was to evaluate at what time of follow-up the radiographic consolidation of the osteotomy was achieved.

SECONDARY OUTCOMES:
AOFAs metatarsophalangeal (MTP)-interphalangeal (IP)- American Orthopaedic Foot & Ankle score. The questionnaire was administered pre-operatively and to some follow-ups in order to evaluate the changes in the patient's clinic. | Preoperative, 90-180-360 days of follow up from the surgery
  Patients completed a clinical evaluation questionnaire (AOFAs metatarsophalangeal (MTP)-interphalangeal (IP)- American Orthopaedic Foot & Ankle score). It is a clinical test commonly used in the scientific literature, which serves to evaluate, in terms of value from 0 to 100, the autonomy, pain, stability, and alignment of the hallux of the patient.
  The questionnaire was collected preoperatively and at 90-180-360 days of follow-up from surgery. No follow-up questionnaires were submitted before 90 days to avoid the influence of post-operative pain.
VAS - Visual Analogue Scale. The questionnaire was administered pre-operatively and to some follow-ups in order to evaluate the changes in the patient's clinic. | Preoperative, 90-180-360 days of follow up from the surgery
  Patients completed a clinical evaluation questionnaire (VAS - Visual Analogue Scale). It is a measurement instrument that tries to measure a characteristic or attitude, for example, the amount of pain that a patient feels ranges across a continuum from none (0) to an extreme amount of pain (10).
  The VAS was collected preoperatively and at 90-180-360 days of follow-up from surgery. No follow-up questionnaires were submitted before 90 days to avoid the influence of post-operative pain.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Russo, MD, Principal Investigator — Istituto Ortopedico Rizzoli